CLINICAL TRIAL: NCT07396454
Title: A Prospective, Single-Arm, Phase II Clinical Study of Radiotherapy Combined With Anlotinib and a Tubulin Inhibitor for the Treatment of HER2-Negative Breast Cancer With Brain Metastases
Brief Title: Study on the Treatment of HER2-negative Breast Cancer Brain Metastases With Radiotherapy Combined With Anlotinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-691
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HER2-Negative Breast Cancer
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Combined with Anlotinib and a Microtubule Inhibitor (Experimental): Based on the size, location and number of brain metastases, an appropriate radiotherapy plan is given. Arloxitin can be used starting from the 1st day after radiotherapy to within 1 week.
  Arloxitin 12 mg, qd (it is recommended to take it before meals and take the medicine at the same time every day), take orally continuously for 2 weeks and then stop for 1 week. A 21-day period constitutes one treatment cycle. During the medication period, if there is a missed dose, if the time from the missed dose to the next dose is less than 12 hours, no additional dose will be given.
  Interventions: Drug: Radiotherapy Combined with Anlotinib and a Microtubule Inhibitor

INTERVENTIONS:
Drug: Radiotherapy Combined with Anlotinib and a Microtubule Inhibitor — Based on the size, location and number of brain metastases, an appropriate radiotherapy plan is given. Arloxitin can be used starting from the 1st day after radiotherapy to within 1 week.
  Arloxitin 12 mg, qd (it is recommended to take it before meals and take the medicine at the same time every day), take orally continuously for 2 weeks and then stop for 1 week. A 21-day period constitutes one treatment cycle. During the medication period, if there is a missed dose, if the time from the missed dose to the next dose is less than 12 hours, no additional dose will be given.

SUMMARY:
Angiogenesis inhibition represents a significant therapeutic target in breast cancer; however, despite its theoretical feasibility, progress in advanced breast cancer has been slow. Currently, there is a lack of prospective data supporting the selection of tyrosine kinase inhibitors (TKIs) in combination with local therapy. This phase II study aims to evaluate the efficacy and safety of stereotactic radiotherapy (SRT) or whole-brain radiotherapy (WBRT) combined with anlotinib in patients with HER2-negative advanced breast cancer and brain metastases.

DETAILED DESCRIPTION:
Angiogenesis inhibition represents a significant therapeutic target in breast cancer; however, despite its theoretical feasibility, progress in advanced breast cancer has been slow. Currently, there is a lack of prospective data supporting the selection of tyrosine kinase inhibitors (TKIs) in combination with local therapy. This phase II study aims to evaluate the efficacy and safety of stereotactic radiotherapy or whole-brain radiotherapy (WBRT) combined with anlotinib in patients with HER2-negative advanced breast cancer and brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 70 years (calculated on the date of informed consent signing).
* Karnofsky Performance Status (KPS) score ≥ 70, or KPS = 60 primarily attributable to neurological symptoms.
* HER2-negative status confirmed by pathology from Jiangsu Provincial Hospital's Pathology Department. HER2 immunohistochemistry (IHC) must be (-) or (1+). Patients with HER2 IHC (2+) must have a negative result on confirmatory fluorescence in situ hybridization (FISH) testing.
* Presence of brain metastases confirmed by contrast-enhanced cranial MRI prior to enrollment. At least one measurable intracranial lesion is required according to RANO-BM criteria.
* If prior anti-tumor therapy (excluding treatments specifically targeting intracranial metastases) has been administered, a washout period of at least 2 weeks is required. Any prior treatment-related toxicities must have resolved to ≤ Grade 2 (CTCAE v3.0; excluding alopecia and hematological toxicities). Concurrent use of bisphosphonates, mannitol, corticosteroids, etc., is permitted during the study. Corticosteroid dosage must have been stable for at least one week prior to enrollment (e.g., dexamethasone ≤ 16 mg/day or equivalent).
* Life expectancy of at least 3 months.
* Adequate organ and hematological function, meeting the following criteria:

  1. Hematology (without transfusion or growth factor support within 14 days):

     * Hemoglobin (Hb) ≥ 80 g/L.
     * Absolute neutrophil count (ANC) ≥ 1.0 × 10⁹/L.
     * Platelet count (PLT) ≥ 50 × 10⁹/L.
  2. Biochemistry:

     * Total bilirubin (TBIL) < 1.5 × upper limit of normal (ULN), or ≤ 3 × ULN in patients with liver metastases.
     * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN, or ≤ 5 × ULN in patients with liver metastases.
     * Serum creatinine (Cr) ≤ 1.5 × ULN or calculated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula).
     * Magnesium ≥ lower limit of normal (LLN).
* Women of childbearing potential must be surgically sterile, postmenopausal, or agree to use highly effective contraception (e.g., oral contraceptives, intrauterine device, sexual abstinence, or barrier methods with spermicide) during the study and for 6 months after the final dose. A negative serum pregnancy test within 7 days prior to enrollment is required for all non-sterile, premenopausal women (positive results must be ruled out as false-positive by ultrasound). Patients must not be breastfeeding.
* Voluntary participation with written informed consent.

Exclusion Criteria:

* Patients with extensive leptomeningeal metastasis or hemorrhagic brain metastases.
* Patients with uncontrolled seizures.
* Patients with any other severe and/or poorly controlled concurrent medical condition that, in the investigator's judgment, prohibits their participation in this clinical study, including but not limited to:

  1. Factors significantly affecting oral drug intake (e.g., inability to swallow, chronic diarrhea, intestinal obstruction).
  2. Known hypersensitivity to anlotinib or any component of the investigational product.
  3. History of immunodeficiency, including HIV positivity, other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
  4. Clinically significant cardiovascular disease (defined as: unstable angina, symptomatic congestive heart failure of New York Heart Association [NYHA] Class ≥ II, uncontrolled severe arrhythmia), or myocardial infarction within 6 months prior to enrollment.
  5. Active or uncontrolled infection requiring systemic treatment within 2 weeks prior to enrollment (excluding simple urinary tract infections or upper respiratory tract infections).
  6. History of concurrent other malignancies, except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patients who are pregnant, breastfeeding, or planning to become pregnant during the treatment period or within 6 months after treatment completion.
* Patients (including female patients and/or their male partners) unwilling to use effective contraception during the treatment period and for 6 months after treatment completion.
* Patients ineligible for contrast-enhanced MRI examinations.
* Patients who have previously received anti-angiogenic TKI therapy and experienced intracranial progression (Note: Patients who received prior anti-angiogenic TKI therapy without subsequent disease progression are eligible. Patients previously treated with anti-angiogenic macromolecular agents, such as bevacizumab, are eligible).
* Patients with a history of other malignancies within the past 5 years or concurrent other malignancies, except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix. (Note: This appears to be a duplicate of criterion 3f. In standard protocols, it is typically listed once.).
* Patients unwilling or unable to comply with scheduled follow-up as required by the study protocol.
* Any other condition assessed by the investigator that may affect the patient's compliance with the protocol or the evaluation of study endpoints, rendering the patient unsuitable for study participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Central nervous system progression-free survival (CNS-PFS) rate | 12months
  According to the RANO-BM (Response Assessment in Neuro-Oncology Brain Metastases) standard, the 12-month central nervous system progression-free survival (CNS-PFS) rate was determined by at least two experienced neuro-radiologists.

SECONDARY OUTCOMES:
Central nervous system progression-free survival (CNS-PFS) | 12months
  It is defined as the time from the start of the study treatment for the subject until the first imaging confirmation of intracranial disease progression (PD) or any cause of death. The assessment of intracranial lesions is based on the RANO-BM standard.
Progression free survival（PFS） | 12months
  It is defined as the time from the start of the study treatment for the subject until the first imaging confirmation of disease progression (PD) or death due to any cause. The assessment of intracranial lesions is based on the RANO-BM criteria, while the assessment of extracranial lesions is based on the RECIST 1.1 criteria.
Overall survival（OS） | 12months
  It is defined as the period from the date of receiving the study treatment to the date of death (due to any cause). For subjects who did not experience death, the analysis will be truncated at the time of confirmed survival.
Objective Response Rate of the Central Nervous System (CNS-ORR) | 12months
  It is defined as the percentage of subjects who achieved complete or partial responses in the central nervous system from the time they began receiving treatment in this study until they left the study group. The assessment is conducted using the RANO-BM criteria.
Karnofsky Performance Status (KPS) score | 12months
  The assessment was conducted using the Karnofsky Performance Status.
Adverse event（AE） | 12months
  AEs are recorded according to the NCI CTCAE 5.0 standard
Simple Mental State Examination (MMSE) score | 12months
  The assessment was conducted using the Mini-Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No